CLINICAL TRIAL: NCT03772106
Title: Effect of Sevoflurane and Propofol on Hepato-splanchnic Pressure and Flow During Hepatobiliary Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2017/0164
Record Dates: First submitted 2018-12-04; First posted 2018-12-11 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: General Anesthesia
Keywords: hepato-splanchnic blood flow
MeSH Terms: interventions — Propofol; Sevoflurane

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group P (Experimental): Group P : Propolipid 1% dose : variable to keep BIS between 40 and 60
  Interventions: Drug: Propofol Fresenius
- Group S (Experimental): Group S : Sevoflurane dose : variable to keep BIS between 40 and 60
  Interventions: Drug: sevorane

INTERVENTIONS:
Drug: Propofol Fresenius — Propolipid 1% : IV
  Arms: Group P
Drug: sevorane — sevorane Quick fill (sevoflurane) : inhalation
  Arms: Group S

SUMMARY:
Blood loss in hepatobiliary surgery is correlated with an increase in postoperative complications (e.g. transfusion related lung injury and tumor recurrence) and reduced longterm survival. To reduce morbidity and mortality in hepatobiliary surgery, modulation of the hepato-splanchnic blood flow and pressure is used. In liver surgery pharmacological modulations are widely used to prevent blood loss. For pharmacological modulation central venous pressure is commonly used to reduce the pressure in the inferior vena cava, however little is known about pharmacological effect on blood flow in the hepatic artery and portal vein. The modulation of the hepato-splanchnic blood flow can also play an important role, not only for prevention of blood loss but also for survival of the organs (e.g. ischemic injury due to low flow).

Volatile anesthetics induce a dose-dependent reduction of the hepato-splanchninc blood flow. Propofol however, increases hepatic blood flow when compared with volatile anesthetics. Pharmacological modulation of hepato-splanchnic bloodflow with anesthetics such as sevoflurane or propofol can play an important role in modulation of ischemia/reperfusion injury and survival of organs.

The aim of the study is to determine and to compare the effect of sevoflurane versus propofol on hepatosplanchnic pressure and hepato-splanchnic blood flow during hepatobiliary surgery.

DETAILED DESCRIPTION:
All patients receive standardized anesthesia care for hepato-biliary surgery according to the existing anesthesia protocol. The type of anaesthesia will be randomized : propolipid (TIV) or sevorane(inhalation).

At designated times, hemodynamic variables will be recorded.

These will include:

* HF (/min)
* CVP (mmHg),
* MAP (mmHg)
* CI (L/min.m2)
* PPV (pulse pressure variation). Hemodynamic measurement will be done using PiCCO catheter.

The hemodynamic measurements will be compared and related to hepato-splanchnic blood flow and pressure measurements performed by the surgeon:

* Flow v. porta
* Flow art. hepatica
* Pressure v. porta
* Pressure v. cava The flow measurements will be done using ultrasound transit time ﬂow measurements TTFM (Medi-Stim AS, Oslo, Norway).

At the same time pressure measurements will be obtained in portal vein and caval vein using a 25-gauge needle which is directly placed in the vein. Both flow and pressure will be simultaneously recorded (VeriQ 4122, Medi-Stim AS, Oslo, Norway). Both measurements will be done during apnea to minimize the effect of ventilation on pressure & flow. Flow values will be expressed in ml per minute, pressure values will be expressed in mmHg.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥ 18 years (Female or Male)
* ASA I - II - III
* Able to comprehend, sign and date the written informed consent document to participate in the clinical trial.
* Scheduled for hepato-biliary surgery.

Exclusion Criteria:

* Allergy for the medication
* Renal insufficiency (SCr > 2 mg/dl)
* Severe heart failure (EF < 25%)
* Hemodynamic instable patients
* Arterial fibrillation
* Sepsis
* BMI > 40
* Severe coagulopathy (INR > 2)
* Thrombocytopenia (< 80 x 10³ /µL)
* History of severe postoperative nausea & vomiting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-06-08 (Actual); Primary Completion 2018-01-27 (Actual); Study Completion 2018-12-04 (Actual)

PRIMARY OUTCOMES:
Change in blood flow in hepatic artery and main portal vein | From randomization until the end of the whipple surgery
  flow/pressure measurements with echo probe and needle

SECONDARY OUTCOMES:
need of inotropic and/or vasopressor support | From start anesthesia until end of anesthesia
  total dose of inotropic and vasopressor medication that were used during surgery
amount of blood loss | From start of surgery until end of surgery
  amount of blood loss at end of surgery
amount of colloids given during surgery | From start of surgery until end of surgery
  total amount of colloids given during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jurgten Van Limmen, MD, Principal Investigator — UZ Ghent
Locations (1):
- University Hospital Ghent, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van Limmen J, Wyffels P, Berrevoet F, Vanlander A, Coeman L, Wouters P, De Hert S, De Baerdemaeker L. Effects of propofol and sevoflurane on hepatic blood flow: a randomized controlled trial. BMC Anesthesiol. 2020 Sep 22;20(1):241. doi: 10.1186/s12871-020-01150-3. PMID 32962657